CLINICAL TRIAL: NCT05259462
Title: Improving Social Isolation and Loneliness Among Children With Physical Disabilities Through Group-Based Online Virtual Reality Gaming
Brief Title: Group-Based Online Virtual Reality Gaming to Improve Mental Health Among Children With Physical Disabilities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Byron Lai, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEDHARS6306
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Disability Physical
Keywords: virtual reality
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Single group pre-to-post design trial that will last 1-year and include 2 waves (n=6 per wave)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-active virtual reality gaming (Experimental): Participants will undergo the intervention.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Participants will utilize low-cost, consumer available head-mounted displays to meet with peers and coaches online. The program will last 4 weeks and include 2 x 1-hour sessions per week of supervised peer-to-peer gaming. The coaches will utilize behavioral change and mindfulness techniques to promote autonomy, competence, and relatedness through a respectful, cohesive, and positive atmosphere. These strategies will be framed by the Self-Determination Theory and learned from the National Center on Health, Physical Activity, and Disability (NCHPAD) mindfulness coaching workshops. Some of the mindfulness-based strategies will include guided breathing focused exercises, body scanning, meditation, and acceptance of social anxiety and shyness

SUMMARY:
COVID-19 has had a negative impact on the mental health of many children with physical disabilities. This project aims to test the potential effects of an online multiplayer virtual reality group-based, active video game program on social isolation and depression and will include a total of 12 children with physical disabilities.

DETAILED DESCRIPTION:
This pilot feasibility study will investigate the potential effects of a revised multiplayer virtual reality exergaming program on depression, socialization, and loneliness among children with physical disabilities. This proposed study will use both quantitative and qualitative research methods, to gain a deep understanding of program benefits and implementation procedures that can be refined for a large clinical trial. The active video game program will last 1-month and include 2 supervised 1-hour sessions per week of group-based gaming. Game sessions will be supervised by 2 research staff who will act as gaming and mindfulness coaches. Outcomes will be measured by self-report questionnaires before and after the program. The program will be completed in two waves (6 people per wave). After the program, participants will undergo a one-on-one semi-structured interview, where they can describe their perceptions of the program.

ELIGIBILITY:
Inclusion Criteria:

* self-reported mobility disability (e.g., use of a mobility device or presence of a mobility impairment)
* access to a Wi-Fi internet connection in the home
* a caregiver to support the child if <18 years of age
* a Facebook account to link to the virtual reality head-mounted display

Exclusion Criteria:

* physically active (defined as >150 minutes/week of moderate-to-vigorous intensity exercise)
* cannot use the arms for exercise or operate the controller buttons using their fingers
* prone to seizures
* complete blindness or deafness
* unable to communicate verbally in English

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in Depression | Changes from baseline (week 0) to post-intervention (week 5)
  Changes in self-reported feelings of depression measured by the Children's Depression Inventory 2 Short Form (CDI-S 2).
Changes in Social Isolation / Loneliness | Changes from baseline (week 0) to post-intervention (week 5)
  Measured by the version 3 of the UCLA Loneliness Scale 20 items (UCLA-20).

SECONDARY OUTCOMES:
Class attendance | Weeks 1 - 4
  Percent of classes attended divided by the total
Exercise volume | Week 0 and Week 5
  Self-reported minutes of exercise per week completed. Measured by the Godin Leisure-Time Exercise Questionnaire (GLTEQ).
Quality of social interactions | Week 5
  A scale measure of how participants felt about the quality of social interactions they had during online virtual reality gameplay. The scale ranges from 1-5, where 5 indicates a very high quality of social interactions and a 1 indicates a very low quality of social interactions.
Perceived enjoyment of the group classes | Week 5
  A scale measure of how enjoyable online group gameplay was. The scale ranges from 1-5, where 5 indicates a very high level of perceived enjoyment with the group classes and a 1 indicates a very low perceived enjoyment with the group classes.
Satisfaction with program delivery | Week 5
  A scale measure of participants' satisfaction with how the classes were conducted. The scale ranges from 1-5, where 5 indicates a very high perceived satisfaction of the program delivery and a 1 indicates a very low perceived satisfaction with the program delivery.
Multiplayer feedback survey | Week 5
  A questionnaire measuring multiplayer playtime (self-reported times played per week), friendship creation (yes/no), and friendship strength (assessed via Likert scale).
Participants Perceptions of Completing the Program | Week 5
  Semi-structured interviews evaluating their perceptions of completing the program, with specific attention to providing more in-depth responses (i.e.,explanations) for each of the 8 outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai B, Young R, Craig M, Chaviano K, Swanson-Kimani E, Wozow C, Davis D, Rimmer JH. Improving Social Isolation and Loneliness Among Adolescents With Physical Disabilities Through Group-Based Virtual Reality Gaming: Feasibility Pre-Post Trial Study. JMIR Form Res. 2023 Dec 6;7:e47630. doi: 10.2196/47630. PMID 38055309
- [Derived] Lai B, Davis D, Young R, Swanson-Kimani E, Wozow C, Chaviano K, Rimmer JH. Group Telegaming Through Immersive Virtual Reality to Improve Mental Health Among Adolescents With Physical Disabilities: Pre- and Posttrial Protocol. JMIR Res Protoc. 2022 Oct 13;11(10):e42651. doi: 10.2196/42651. PMID 36194864